CLINICAL TRIAL: NCT01736111
Title: Text Messaging for Weight Loss in Primary Care Patients
Brief Title: Text Messaging for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Kevin Hwang, MD, Assistant Professor - Internal Medicine, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-12-0571
Record Dates: First submitted 2012-11-07; First posted 2012-11-29 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Obesity
Keywords: obesity; weight loss; text message
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Personal feedback (Experimental): This arm will receive all intervention components of Active Comparator group, plus the following:
  1. Text messages to prompt participant to reply with self-monitoring entries
  2. Human coach uses system to send personalized text messages with feedback on self-monitoring entries
  Interventions: Behavioral: Personal feedback
- One Way Text (Active Comparator): 1. Printed handouts from the "Aim for a Healthy Weight" booklet, which is published by National Heart, Lung, and Blood Institute and is frequently included in control conditions in primary care-based weight loss studies.
     Other handouts will discuss the use of prepackaged foods as well as setting goals for calorie intake, physical activity, and weight loss.
  2. One to three text messages per week, based on topics from "Aim for a Healthy Weight" and other sources. The text messages will be pre-scheduled, automated, non-tailored, and "one-way" (no reply will be requested). The total dose of contact will be low because each text message is limited to 160 characters. The condition is comparable in intensity to control conditions in other weight loss trials in the primary care setting.
  3. Usual medical care from the PCP.
  4. Education on symptoms of hypoglycemia, hypotension, and cardiovascular disease, with instructions to contact their PCP in the event of those symptoms.
  Interventions: Behavioral: one way text

INTERVENTIONS:
Behavioral: one way text
  Arms: One Way Text
Behavioral: Personal feedback
  Arms: Personal feedback

SUMMARY:
Overweight and obese adults recruited from the primary care setting (n=150) will be enrolled in a 6-month randomized trial of the INTERVENTION versus CONTROL. Both groups will receive usual medical care, printed materials, and educational text messages. The INTERVENTION group will also receive personalized coaching and feedback, as well as peer support, via text message.

The investigators hypothesize that compared to those in the Control group, patients in the Intervention group will lose more weight and demonstrate more favorable changes in fruit and vegetable intake, exercise, and social support for weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Approved to participate by PCP (Patients with diabetes, hypertension, or dyslipidemia will be eligible if approved by their PCP)
* Age ≥ 21 years
* Body mass index (BMI) 25 to 45 kg/m2 and weight ≤ 400 pounds
* Goal of losing weight (not just maintain weight)
* Willing to change diet, physical activity in order to lose weight.
* Currently uses text messaging in English on mobile phone
* Willing to use send and receive text messages for this study without direct compensation for cost of messages (general compensation for study participation will be provided)
* Have a scale at home for self-monitoring weight
* Fluent in English (speak, read, write)
* Commit to return for follow-up weight at 6 months regardless of amount of weight lost

Exclusion Criteria:

* Involuntary or voluntary weight loss of ≥ 5% body weight in previous 6 months
* Participating in research project involving weight loss, exercise, or dietary modification in the previous 6 months
* Any of the following medical conditions which could affect weight or for which weight loss is contraindicated

  * End-stage liver disease
  * End-stage kidney disease
  * Cancer within previous 2 years (except non-melanoma skin cancer)
* Myocardial infarction, stroke, or transient ischemic attack within previous 6 months
* Unstable angina
* Severe arthritis or other medical conditions which would prevent brisk walking
* Schizophrenia
* Hospitalization for psychiatric problems during the prior 12 months.
* Current use or anticipated future use (during 6 month study) of medications that could cause weight loss:

  * phentermine
  * orlistat (prescription Xenical or OTC Alli)
  * topiramate
  * buprioprion
  * exenatide (Byetta)
  * liraglutide (Victoza)
* Prior bariatric surgery or plans for bariatric surgery in next 6 months
* Pregnant or breast feeding within the previous 6 months
* Planning to become pregnant in next 6 months
* Consumes > 14 alcoholic drinks per week
* Current use of illicit drugs
* Planning to move out of the area in the next 6 months
* Another member of household or a close contact is participating in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in weight from baseline | baseline and 6 months
  Weight in a lightweight hospital gown with no shoes (calibrated digital scale)

SECONDARY OUTCOMES:
Change in diet measured by Fruit and Vegetable Screener (NCI) | baseline and 6 months
Change in physical activity as measured by Paffenbarger physical activity questionnaire | baseline and 6 months
Change in social support as measured by Weight Management Support Inventory | baseline and 6 months
  A validated questionnaire with 4 domains of social support for weight control (emotional, instrumental, informational, and appraisal)
Change in executive function as measured by Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) | baseline and 6 months
  Measures the individual's self-rated executive functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin O. Hwang, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- UT Physicians - Internal Medicine, Houston, Texas, United States